CLINICAL TRIAL: NCT01374295
Title: Video Assisted Informed Consent for Lortab to Improve Patient Satisfaction and Knowledge: A Randomized Control Study
Brief Title: Video Assisted Informed Consent for Lortab to Improve Patient Satisfaction and Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Wayne Triner, Professor Dept. of Emergency Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2981; Lortab
Record Dates: First submitted 2011-06-07; First posted 2011-06-15 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2011-06

CONDITIONS: Non-critical Emergency Room Patients Receiving Lortab Medication or Prescription During Their Emergency Room Visit
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- video (Experimental): If randomized to this arm patient watches a 3 minute video
  Interventions: Other: video
- standard education (Active Comparator): If randomized to this arm patient receives standard verbal education from healthcare provider.
  Interventions: Other: standard education

INTERVENTIONS:
Other: video — watch a 3 minute video
  Arms: video
Other: standard education — Receives standard verbal education from healthcare provider
  Arms: standard education

SUMMARY:
In order to compare two different forms of patient education; patients who receive Lortab medication or prescription during their ED visit are randomized to receive either standard patient education (from healthcare provider) or video assisted education. After education, patient completes a survey, estimated to take 5 minutes to complete.

DETAILED DESCRIPTION:
The purpose of this study is to compare different methods of teaching patients about their prescription medicines. It is possible that certain teaching methods are better than others at educating patients.

Patients who receive Lortab medication or prescription during their ED visit and agree to the study are randomized to receive either standard patient education (from healthcare provider) or watch a 3 minute video. After the medication teaching has been provided the patient is given the medicine and a asked to complete a ten-question survey. This takes approximately five minutes and asks the patient to rate the quality of the information received.

ELIGIBILITY:
Inclusion Criteria:

* non-critical emergency room patients being prescribed Lortab
* age 18 year or older

Exclusion Criteria:

* emergency room patients not receiving Lortab as their first prescribed medication
* age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction and knowledge | survey is completed immediately after education, estimated time to complete survey is 5 minutes
  comparison of patient completed survey following education via standard format or 3 minute video

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States